CLINICAL TRIAL: NCT02029768
Title: Gender Disparity in Burn Injury Survival
Status: Terminated | Type: Observational
Why Stopped: Could not reach recruitment goal
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Laura W. Bush Institute for Women's Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: L14-029
Record Dates: First submitted 2014-01-02; First posted 2014-01-08 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Obesity; Burn Injury
Keywords: outcome
MeSH Terms: conditions — Obesity; Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples Without DNA — Serum samples to be used for cytokine measurements
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with burn injury
- Men with burn injury

SUMMARY:
Hypothesis 1: A quantifiable difference in inflammatory cytokines exist in women with burn injury and this correlates with clinical markers of outcome

Hypothesis 2: The amount of adipose tissue contributes to the severity of cellular immune response (CMI) dysregulation in response to burn injury

Skin-fold caliper measurements will be taken on consented patients (both male and female) to determine body fat percentage. Serum samples will be obtained from these patients. The level of inflammatory cytokines in the serum will be measured to determine if there is a link between body fat percentage, pro-inflammatory cytokines and the ability of women to survive burn injury.

DETAILED DESCRIPTION:
Consented patients admitted to University Medical Center with greater than 15% total body surface area burns will participate in this study. A skin-fold caliper measurement will be performed to determine body fat percentage. Serum samples will be obtained and assayed for inflammatory cytokines to establish whether or not a link between obesity in women and pro-inflammatory cytokines exists. If so, obesity may be a factor which contributes to the gender disparity in burn wound survival.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 65 years
* Admitted to University Medical Center with greater than 15% total body surface area burns
* Able to provide informed consent or has authorized representative to give informed consent

Exclusion Criteria:

* Prisoners or pregnant women
* Individuals with injuries that preclude taking caliper measurements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be derived from adult patients admitted to the University Medical Center with greater than 15% total body surface area burns
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Inflammatory cytokine levels | 72 hours post admission until patient discharge
  We will measure inflammatory cytokine levels and determine if elevated cytokine levels are linked to obesity and ultimately burn injury survival

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center/University Medical Center, Lubbock, Texas, United States